CLINICAL TRIAL: NCT02224599
Title: Phase I/II Study of Low-Dose Cyclophosphamide, Tumor Associated Peptide Antigen-Pulsed Dendritic Cell Therapy and Imiquimod, in Patients With Progressive and/or Refractory Solid Malignancies
Brief Title: Cyclophosphamide, TAPA-Pulsed Dendritic Cell Therapy and Imiquimod in Progressive and/or Refractory Solid Malignancies
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to terminate study due to poor accrual
Sponsor: Kiromic BioPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KIROVAX-003
Record Dates: First submitted 2014-08-11; First posted 2014-08-25 (Estimated); Results first posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-03

CONDITIONS: Progressive Solid Malignancies; Refractory Solid Malignancies; Cancer
Keywords: Immunotherapy; TAPA-Pulsed Dendritic Cell Therapy; Dendritic Cell Therapy
MeSH Terms: conditions — Neoplasms | interventions — Cyclophosphamide; Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CYP, TAPA-pulsed DC vaccine, Imiquimod (Experimental): TAPA-Pulsed DC Vaccine Cyclophosphamide Pill Imiquimod Topical Cream
  Interventions: Biological: TAPA-pulsed DC vaccine; Drug: Cyclophosphamide Pill; Drug: Imiquimod Topical Cream

INTERVENTIONS:
Biological: TAPA-pulsed DC vaccine — Subjects will given the vaccine which contains 1 x 10^7 TAPA-pulsed dendritic cells and is administered ID. A total of three (3) cycles therapy will be administered weekly.
Drug: Cyclophosphamide Pill — Subjects will be given low-dose cyclophosphamide by mouth for 5 days starting 5 to 7 days prior to the vaccine cycle.
  Other Names: Cytoxan®, Neosar®
Drug: Imiquimod Topical Cream — Topical Imiquimod Cream will be applied after vaccination.
  Other Names: Aldara Cream, Zyclara

SUMMARY:
Patients diagnosed with progressive and/or refractory solid malignancies, who have failed conventional therapy, and have no available, potentially curative therapeutic options, will be candidates for this Phase I/II study. Following confirmation of disease progression and/or refractoriness, eligible patients who agree to participate and sign an informed consent form will have their tumor cells/tissues and/or blood analyzed for the expression of a specific panel of Tumor Associated Peptide Antigens (TAPAs), including Sp17, ropporin, AKAP-4, PTTG1, Span-xb, Her-2/neu, HM1.24, NY-ESO-1 and MAGE-1.

DETAILED DESCRIPTION:
For patients whose tumors express one (1) or more of these TAPAs (Sp17, ropporin, AKAP-4, PTTG1, Span-xb, Her-2/neu, HM1.24, NY-ESO-1 and MAGE-1), whole blood will be obtained by phlebotomy and/or leukapheresis performed for generation of autologous DCs. Patient's DCs will be generated in Kiromic's Cell Processing GMP facility, according to established Standard Operating Procedures, and activated by pulsing/loading them with the TAPA(s) relevant for each particular patient. Patients will receive five (5) days of low-dose cyclophosphamide 5 to 7 days prior to each vaccination with TAPA-pulsed DCs to decrease Treg activity. Patients will also receive a single dose of topical Imiquimod cream after each vaccination. TAPA-pulsed DCs will be administered at a fixed dose of up to 1 X 107 DCs. DC vaccination schedule will be weekly via intradermal (ID) injections for a total of 3 vaccinations. Topical Imiquimod cream will also be administered once after the vaccination. Patients will be followed on a weekly basis (or more frequently if required) to evaluate treatment-related toxicity. Immune efficacy and anti-tumor responses will be evaluated per protocol specifications. Continuation and stopping rules for the study will be defined based on toxicity/tolerability (Phase I) and immune efficacy (Phase II).

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent.
2. Patients with histologically proven progressive and/or refractory SM, s/p conventional salvage therapy, completed at least 3 weeks prior to study vaccination, will be eligible for enrollment.
3. Expression of one (1) or more of the following TAPAs: Sp17, AKAP-4, Ropporin, PTTG-1, Span-xb, Her-2/neu, HM1.24, NY-ESO-1 and MAGE-1, by either RT-PCR and/or immunocytochemistry, Western blotting or ELISA, in neoplastic cells and/or blood. For HER-2/neu expression, positive FISH results are acceptable.
4. Presence of measurable or evaluable disease.
5. Patients must not have any active infectious process.
6. Patients must not have a history of HIV, or active Hepatitis A, B, and C.
7. Patients must not be receiving active immunosuppressive therapy.
8. Patients must have discontinued systemic cytotoxic or radiation therapy at least three (3) weeks prior to vaccination and toxicities from previous therapies must be grade 1 or less. all other FDA approved forms of antineoplastic therapy are allowed such as immunotherapy, targeted therapies, or hormonal therapies (67, 68)
9. Patients may not have any known allergy to CYP and/or Imiquimod.
10. Patients must be willing to provide at least 250 mL, and up to 500 mL, of whole blood obtained by phlebotomy and/or consent to leukapheresis for DC generation.
11. Adequate renal and hepatic function (creatinine ≤ 2.0 mg/dl, bilirubin ≤ 2.0 mg/dl, AST and ALT ≤ 4X upper limit of normal range).
12. Adequate hematologic function (Platelets ≥ 60,000/mm3, lymphocytes ≥ 1,000 mm3, neutrophils ≥ 750/mm3, hemoglobin ≥ 9.0 g/dl).
13. Karnofsky performance status ≥ 70%.
14. Expected survival ≥ 6 months.
15. Either a female or male of reproductive capacity wishing to participate in this study must be using, or agree to use, one or more types of birth control during the entire study and for 3 months after completing the study. Birth control methods may include condoms, diaphragms, birth control pills, spermicidal gels or foams, anti-gonadotropin injections, intrauterine devices (IUD), surgical sterilization, or subcutaneous implants. Another choice is for a subject's sexual partner to use one of these birth control methods. Women of reproductive capacity will be required to undergo a urine pregnancy test before completion of the post-screening informed consent process.

Exclusion Criteria:

1. Patients without confirmed progressive and/or refractory SM using standard RECIST criteria.
2. Patients without measurable or evaluable disease.
3. Patients receiving cytotoxic therapy or radiation therapy, within three (3) weeks of vaccination.
4. Active immunosuppressive therapy, including non-physiologic systemic steroids (excluding topical, intraocular, inhaled, and intranasal steroids) for any other condition.
5. Persistent fever (>24 hours) documented by repeated measurement or active, uncontrolled infection within 4 weeks of enrollment.
6. Active ischemic heart disease or history of myocardial infarction within six months.
7. Active autoimmune disease, including, but not limited to, Systemic Lupus Erythematosus (SLE), Multiple Sclerosis (MS), Ankylosing Spondylitis (AS), Inflammatory Bowel Disease (IBD) and Rheumatoid Arthritis (RA).
8. Pregnancy or breast feeding.
9. Active second invasive malignancy, other than basal cell carcinoma of the skin.
10. Life expectancy of less than 6 months.
11. Patients with contraindications to CYP and/or Imiquimod.
12. Patients who have received organ transplants.
13. Patients with psychological or geographic conditions that prevent adequate follow- up or compliance with the study protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-07-28 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Tolcher, MD, Principal Investigator — NEXT Oncology
Locations (1):
- San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CYP, TAPA-pulsed DC Vaccine, Imiquimod
Started | 3
Completed | 1
Not Completed | 2
Not completed — Physician Decision | 1
Not completed — Progression of Disease | 1

BASELINE CHARACTERISTICS:
Arm/Group | CYP, TAPA-pulsed DC Vaccine, Imiquimod
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.33 (18.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Adverse Events Due to Administration of TAPA-Pulse DC Vaccine
Description: Grade, causality, start/stop dates (duration), resolutions for adverse events will be monitored and recorded.
Time Frame: Continuous for 45 days after the first dose.
Population: Enrollment was terminated
Arm/Group | CYP, TAPA-pulsed DC Vaccine, Imiquimod
Number analyzed (Participants) | 0

2. Secondary Outcome: Immune Response
Description: The response of T-cells present in the peripheral blood mononuclear cells (PBMCs) population to the peptides used to pulse a patient's dendritic cell vaccine is evaluated by measuring the expression of Th1/CTL-type cytokines (IFN-γ and/or TNF-α and/or IL-17) by a standard ELI-Spot assay using 500,000 PBMCs per experimental replicate and a minimum of 3 experimental replicates for each stimulation. The results are expressed as the average number of spots obtained from the stimulation of 500,000 PBMCs
Time Frame: Days -7, 22 and 45
Population: Enrollment was teriminated.
Arm/Group | CYP, TAPA-pulsed DC Vaccine, Imiquimod
Number analyzed (Participants) | 0

3. Secondary Outcome: Positive DTH Skin Tests With Relevant TAPA
Description: DTH skin test will be performed on subject's forearm or within 5 cm from the site of prior DC vaccination, if possible
Time Frame: Days -7, 22 and 45
Population: Enrollment was terminated
Arm/Group | CYP, TAPA-pulsed DC Vaccine, Imiquimod
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 8 months
Description: Enrollment was terminated
Arm/Group | CYP, TAPA-pulsed DC Vaccine, Imiquimod
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT02224599/Prot_SAP_001.pdf
  • Informed Consent Form (2018-10-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT02224599/ICF_002.pdf